CLINICAL TRIAL: NCT05454800
Title: Effects of Physical Activity Counseling in Addition to Scoliosis-Specific Corrective Exercises in Patients With Adolescent Idiopathic Scoliosis
Brief Title: Effects of Physical Activity Counseling in Patients With Adolescent Idiopathic Scoliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Pelin Vural, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-FTR9174
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Scoliosis; Adolescent Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scoliosis Specific Corrective Exercises and Physical Activity Counseling (Experimental): Individuals with AIS in this group, in accordance with the Schroth classification, individually planned, aimed at correcting and stabilizing the spine in three dimensions, an exercise program will be applied in 45-60 minutes sessions, 2 days a week, for 8 weeks, a total of 16 sessions. In addition to corrective exercises specific to scoliosis, physical activity counseling will also be given.
  Interventions: Other: Scoliosis Specific Corrective Exercises and Physical Activity Counseling
- Scoliosis Specific Corrective Exercises (Experimental): Individuals with AIS in this group, in accordance with the Schroth classification, individually planned, aimed at correcting and stabilizing the spine in three dimensions, an exercise program will be applied in 45-60 minutes sessions, 2 days a week, for 8 weeks, a total of 16 sessions.
  Interventions: Other: Scoliosis Specific Corrective Exercises

INTERVENTIONS:
Other: Scoliosis Specific Corrective Exercises and Physical Activity Counseling — Scoliosis specific corrective exercises and physical activity counseling
  Arms: Scoliosis Specific Corrective Exercises and Physical Activity Counseling
Other: Scoliosis Specific Corrective Exercises — Only scoliosis specific corrective exercises
  Arms: Scoliosis Specific Corrective Exercises

SUMMARY:
Scoliosis is a three-dimensional deformity of the spine of unknown etiology and is clinically defined as 10° or more lateral curvature of the spine. Although there are different types of scoliosis, the most common type is adolescent idiopathic scoliosis (AIS), which starts at the age of 10. AIS can affect body alignment, spine and soft tissues and cause physical problems such as postural disorder, cosmetic trunk deformity, decreased flexibility of the spinal column, changes in spinal muscle characteristics, and back pain. The aim of our study is to examine the effects of physical activity counseling on physical activity level and posture, perception of deformity and quality of life in patients with AIS.

DETAILED DESCRIPTION:
AIS is the most common spinal deformity seen by primary care physicians, pediatricians, and spinal surgeons. The primary goal in the conservative treatment of scoliosis in adolescents is to prevent the progression of the curvature and secondary problems associated with spinal deformity and ultimately to eliminate the need for surgery. For this reason, scoliosis-specific corrective exercise therapy given by a physiotherapist is recommended for patients with AIS. However, while this treatment is effective to the gold standard on spine and posture, its effect on physical activity is not known exactly. The aim of this study is to examine the effect of physical activity counseling on physical activity level and posture, perception of deformity and quality of life in individuals with AIS who are given physical activity counseling in addition to scoliosis-specific corrective exercises. Individuals with AIS in both groups, in accordance with the Schroth classification, individually planned exercise program aimed at correcting and stabilizing the spine in three dimensions, in the form of 45-60 minutes sessions, 2 days a week for 8 weeks, a total of 16 sessions. Group 1 will be given physical activity counseling as well as scoliosis-specific corrective exercises. Physical activity counseling will be done face-to-face, and one-on-one interviews will be provided with each participant. Each meeting will last approximately 20-30 minutes and individuals will be encouraged to participate in more physical activity by providing alternative solutions on their physical activity habits, what they like to do or how they can access activities.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Idiopathic Scoliosis by an orthopedic specialist
* Cobb angle determined on anteroposterior radiograph is 10 - 45 degrees

Exclusion Criteria:

* Having mental problem, rheumatological, neuromuscular, cardiovascular, pulmonary disease
* Any treatment approach for scoliosis in the last six months
* Having any orthopedic problems that may affect their participation in exercise and/or physical activity
* Having a regular exercise habit

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
The Physical Activity Questionnaire for Older Children (PAQ-C) (The change between the baseline value and the post-follow-up value will be evaluated) | Baseline, end of weeks 8 and six month follow up
  PAQ-C was developed to evaluate the physical activity levels of children aged 8-14 years in the last 7 days. 9 out of 10 items that make up the scale are used to calculate activity scores. The 10th item evaluates whether the child is able to engage in normal activities due to being sick in the previous week or for another reason, but item 10 is not included in the calculation of the activity score. The overall MFAQ score is the average of the scores of 9 items and ranges from 1 to 5. On average, 1 point indicates low physical activity level, and 5 points indicate high physical activity level.
Physical Activity Questionnaire for Adolescents (PAQ-A) (The change between the baseline value and the post-follow-up value will be evaluated) | Baseline, end of weeks 8 and six month follow up
  PAQ-A was developed to evaluate the physical activity levels of adolescents aged 14-20 in the last 7 days. 8 out of 9 items that make up the scale are used to calculate activity scores. Item 9 assesses whether the child is able to engage in normal activities due to illness or other reasons in the previous week, but item 9 is not included in the calculation of the activity score. The overall MFAQ score is the average of the scores of 8 items and ranges from 1 to 5. On average, 1 point indicates low physical activity level, and 5 points indicate high physical activity level.
One-Week Step Count Measurement with Pedometer for Physical Activity Assessment (The change between the baseline value and the post-follow-up value will be evaluated) | Baseline, end of weeks 8 and six month follow up
  It is one of the objective methods used to evaluate physical activity. It is used to record the number of steps taken. The estimated step length is entered into the device and recorded as a step when the vertical oscillation of the body exceeds a certain threshold value. In our study, the number of steps taken by the participants during a week before and after treatment will be calculated and recorded. Higher scores better outcomes.

SECONDARY OUTCOMES:
POsterior Trunk Symmetry Index (POTSI) (The change between the baseline value and the post-follow-up value will be evaluated) | Baseline, end of weeks 8 and six month follow up
  POTSI is defined as the sum of six indices, three frontal plane asymmetry indices and three frontal plane height difference indices, in the patient's anterior and posterior photographs. Calculation is made by placing indices into the formula. While zero represents full symmetry, as the score increases, the asymmetry also increases (Stolinski et al. 2012; Patias et al. 2010). In our study, "SCODIAC" (SCOliotic DIAgnostiCs) computer program will be used for PGAI and AGAI calculations. While zero represents complete symmetry, as the score increases, so does the asymmetry.
Anterior Trunk Symmetry Index (ATSI) (The change between the baseline value and the post-follow-up value will be evaluated) | Baseline, end of weeks 8 and six month follow up
  ATSI (PGAI) is defined as the sum of six indices, three frontal plane asymmetry indices and three frontal plane height difference indices, in the patient's anterior and posterior photographs. Calculation is made by placing indices into the formula. While zero represents full symmetry, as the score increases, the asymmetry also increases (Stolinski et al. 2012; Patias et al. 2010). In our study, "SCODIAC" (SCOliotic DIAgnostiCs) computer program will be used for PGAI and AGAI calculations. While zero represents complete symmetry, as the score increases, so does the asymmetry.
The Walter Reed Visual Assessment Scale (WRVAS) (The change between the baseline value and the post-follow-up value will be evaluated) | Baseline, end of weeks 8 and six month follow up
  WRVAS is an easy-to-use and scoring scale that allows to understand the visual change caused by scoliosis. In WRVAS, which correlates with the degree of curvature and has high internal consistency, treatment results are evaluated under seven headings. Each deformity is scored from 1 to 5 on the scale. In our study, this scale will be filled by the physiotherapist and the individual with AIS, and the difference (dWRVAS) between the WRVAS scores of the physiotherapist and the individual with AIS will be noted. The decrease in the difference will be evaluated as an improvement in the perception of deformity. High scores indicate increased deformity.
The Scoliosis Research Society-22 Questionnaire (SRS-22) (The change between the baseline value and the post-follow-up value will be evaluated) | Baseline, end of weeks 8 and six month follow up
  SRS-22 is a questionnaire designed by the Scoliosis Research Society (SRS) specifically for patients with spinal deformity. This questionnaire, which consists of 5 main titles, includes questions about pain, body image, function, mental health and satisfaction with treatment. The score for each item ranges from zero (worst) to five (best). Scores in the sections can be obtained separately by dividing the score received from each section by the number of questions in the relevant section, and the total score can be obtained by adding the scores obtained from all questions and dividing them by the total number of questions. As a result of scoring, a high score indicates an increase in quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Zengin Alpozgen, PhD, Study Chair — Istanbul University-Cerrahpaşa Faculty of Health Sciences; Ugur Ovacık, MSc., Study Chair — Istanbul University-Cerrahpaşa, Graduate Education Institute; Elcin Akyurek, MSc., Study Chair — Istanbul University-Cerrahpaşa, Graduate Education Institute; Turgut Akgul, MD, Study Chair — Istanbul University Faculty of Medicine; Pelin Vural, MSc., Study Chair — Istanbul University-Cerrahpasa Institute of Postgraduate Education
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Patias P, Grivas TB, Kaspiris A, Aggouris C, Drakoutos E. A review of the trunk surface metrics used as Scoliosis and other deformities evaluation indices. Scoliosis. 2010 Jun 29;5:12. doi: 10.1186/1748-7161-5-12. PMID 20584340
- [Result] Stolinski L, Kotwicki T, Czaprowski D, Chowanska J, Suzuki N. Analysis of the Anterior Trunk Symmetry Index (ATSI). Preliminary report. Stud Health Technol Inform. 2012;176:242-6. PMID 22744500